CLINICAL TRIAL: NCT02126059
Title: The Health Effects of Cognitive Stimulation, Reminiscence, and Aroma-massage Complementary Interventions on Different Behavior Patterns of Patients With Dementia: Comparative and Longitudinal Research
Brief Title: Complementary Interventions on Patients With Dementia: Comparative and Longitudinal Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: Sellin127
Record Dates: First submitted 2014-04-21; First posted 2014-04-29 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Dementia
Keywords: dementia; behavioral and psychological symptoms; quality of life
MeSH Terms: conditions — Dementia; Behavior

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cognitive stimulation (Experimental): One cognitive stimulation session per week for a continuous 10 weeks, each session contains 50 minutes, totally 10 session topics related to cognitive stimulation.
  Interventions: Behavioral: Reminiscence
- Aroma-massage (Experimental): One hand and shoulder massage session per week for a continuous 10 weeks, each session contains 30 minutes, totally 10 session massage.
  Interventions: Behavioral: Cognitive stimulation
- reminiscence (Experimental): One reminiscence session per week for a continuous 10 weeks, each session contains 50 minutes, totally 10 session topics related to reminiscence.
  Interventions: Behavioral: Aroma-massage
- Control (No Intervention): Control group remain regular activities

INTERVENTIONS:
Behavioral: Reminiscence — The 10 session topics include "Happy to seeing you", "Childhood stories", "Food flavor", "Our old songs", "Festival", "My family", "My Carrier", "Unforgettable events", "My home", and "My award".
  small group intervention (8-12 per group), expected total number of group is 5.
  Other Names: Reminiscence complementary therapy
  Arms: Cognitive stimulation
Behavioral: Cognitive stimulation — The 10 session topics include "psycial activities", "sound", "face", "food", "word association", "number and games", "being creative", "categorizing objects", "orientation", and "team qiuz".
  small group intervention (8-12 per group), total number of group is 5.
  Arms: Aroma-massage
Behavioral: Aroma-massage — Researcher will conduct hand and arm massage to a patient, once a week, each time session for 30 mins with natural tested and safe aroma-essential oil.
  Arms: reminiscence

SUMMARY:
Cognitive function, behavioral and psychological symptoms, and quality of life will improve after administration of cognitive stimulation therapy, reminiscence therapy, and aroma-massage therapy in patients with dementia.

DETAILED DESCRIPTION:
This study will base on the pattern of behavioral and psychological symptoms of dementia, to verify and compare the effectiveness of the three non-pharmacological complementary interventions, cognitive stimulation therapy, reminiscence therapy, and aroma-massage therapy on patients' cognitive function, behavior and psychological symptoms, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* been diagnosed with dementia (all stages) or MMSE below 23 for high school educated and 17 for less than high school education
* able to communicate verbally or nonverbally
* able to understand short sentences
* can sit for at least 50 mins.

Exclusion Criteria:

* no hospitalization within the past two weeks
* not under severe acute illness
* no psychiatric disorders.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
behavioral and psychological symptoms of dementia | 2 years
  To examine if patients' behavioral and psychological symptoms decrease after the intervention.
  Chinese version of Cohen-Mansfield Agitation Inventory (CMAI) will be used to measure this outcome.
  Data will be analyzed through GLM repeated measure-GEE.

SECONDARY OUTCOMES:
quality of life | 2 years
  To examine if patients' quality of life improve after the intervention. WHO Quality of Life-brief Taiwanese version (WHOQOL-BREF) will be used to measure this outcome.
  Data will be analyzed through GLM-repeated measure-GEE.

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Jy Wang, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University Dementia center, Tainan, Taiwan

REFERENCES:
- [Derived] Ball EL, Owen-Booth B, Gray A, Shenkin SD, Hewitt J, McCleery J. Aromatherapy for dementia. Cochrane Database Syst Rev. 2020 Aug 19;8(8):CD003150. doi: 10.1002/14651858.CD003150.pub3. PMID 32813272